CLINICAL TRIAL: NCT07360613
Title: A Pilot Evaluation of the Effectiveness and Economic Impact of a Multi-Technology Rehabilitation Programme for Sub-acute Stroke Patients
Brief Title: Effect of Technology Enriched Rehabilitation After Stroke
Acronym: EFTERS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Strathclyde (Other)
Collaborators: NHS Lanarkshire (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UEC/Kerr_IRAS_359369
Record Dates: First submitted 2025-11-26; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Rehabilitation
Keywords: Rehabilitation; Technology; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Baselines measures of mobility (Primary: Rivermead Mobility Index) before the intervention. Intervention a rehabilitation programme delivered through technology (VR, Treadmills, hand trainers, power assisted exercise). Measures of Mobility repeated immediately before hospital discharge.
Masking Description: No masking is used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Technology Enriched Rehabilitation (Experimental): The intervention is a rehabilitation programme delivered entirely through technology, including virtual reality (immersed and non-immersed), treadmills, weight suspension and movement resistance, and power assistance equipment located in a gym-like space located on an acute stroke unit.
  Individual programs are designed and reviewed by a physiotherapist using principles of intensity, feedback, cognitive engagement, and aerobic activity to address the goals identified by the participant and scores from outcome measures at baseline. Supervision is provided by rehabilitation assistants Participants attend according to their tolerance (assessed by clinical team) up to 2 hours per day until discharged home.
  Interventions: Other: Technology Enriched Rehabilitation

INTERVENTIONS:
Other: Technology Enriched Rehabilitation — The intervention is a rehabilitation programme delivered entirely through technology, including virtual reality (immersed and non-immersed), treadmills, weight suspension and movement resistance, and power assistance equipment located in a gym-like space on an acute stroke unit (NHS Lanarkshire). Individual programs are designed and reviewed by a physiotherapist using principles of intensity, feedback, cognitive engagement, and aerobic activity to address the goals identified by the participant and scores from outcome measures at baseline. Attendance at the gym is supervised and assisted by rehabilitation support workers. Participants can attend daily for 2 hours maximum until discharge, according to their tolerance and judgement of the clinical ward team.

SUMMARY:
The Biomedical Engineering Dept, University of Strathclyde, co-creates rehabilitation technology. In 2023-2024 a clinical study (NCT06787768) was conducted to understand the feasibility of a multi-technology approach to rehabilitation early after stroke. This was successful and leads to the next phase which is to gather preliminary evidence of the effectiveness of this approach by monitoring change in the mobility of patients who receive this intervention compared with usual care which will be gathered through a data linkage project (tracking the outcomes from matched patients from other parts of Scotland who receive usual care).

DETAILED DESCRIPTION:
Rationale A well-established multi-disciplinary research group at the University of Strathclyde (UoS) Biomedical Engineering department have developed and tested a multi-technology rehabilitation model as a solution to the gap between clinical need and current provision. The technology enriched rehabilitation model has been tested under controlled conditions with chronic stroke survivors (at least one-year post stroke) and shown to be feasible with preliminary evidence of efficacy. The model has since been tested on acute/sub-acute stroke patients in an NHS stroke unit and found to be feasible and clinically acceptable with early evidence of an increased rehabilitation dose. This early stroke population has greater potential for recovery as the brain is more receptive to recovery through structural changes to neural pathways (neuroplasticity), therefore delivering higher intensity rehabilitation is therefore more critical at this phase of rehabilitation.

Funding has now been secured to progress this work by gathering evidence on the effectiveness of this approach in recovery mobility (walking, balance and) as well as gathering preliminary evidence of cost effectiveness (healthcare use).

Overall aim To determine whether early, technology-based rehabilitation after stroke improves mobility compared with usual care, using a virtual control group from national linked data, and to identify factors that influence recovery and assess economic benefit.

Specific questions;

1. In sub-acute stroke, does technology-enhanced rehabilitation improve mobility (mRMI) versus a virtual usual-care control identified via a data linkage study, 3 and 6 months after stroke?
2. What is the relationship between delivered dose (hours of rehabilitation) and outcome?
3. Which baseline factors influence outcomes?
4. What are the potential economic benefits of the technology-based rehabilitation programme compared with usual care, based on differences in healthcare and social care resource use and patient outcomes, using national linked data?

Outcome measures The primary variable for comparison will be the modified Rivermead Mobility Index (mRMI) which is a standard measure of mobility routinely used in the NHS, including NHS Lanarkshire. In addition to this the research team will carry out the following tests before the intervention and before discharge.

Measures of motor recovery:

10mwt, five times sit to stand, short version of the BERG Balance Scale, Timed up and Go test, Action Research Arm Test

Health economic measures:

Length of initial stay, Hospital readmissions, stroke recurrence, mortality, Prescription use, GP visits, Level of paid social care STUDY DESIGN and METHODS of DATA COLLECTION AND DATA ANALYIS This is a phase 2, Pre-post design with a non-equivalent virtual control group (VCG) from data linkage study in line with Medical Research Council recommendations for development of a complex intervention.

* Inpatients on the stroke unit at University Hospital Wishaw will be assessed for broad eligibility by the NHS multidisciplinary team using the inclusion/exclusion criteria.
* Patients who have been identified as medically fit for rehabilitation and who fit the criteria for the study shall be highlighted to the research assistant by the NHS medical/therapy team. The researcher shall then check with the relevant members of the multi-disciplinary team that all inclusion/exclusion criteria are met before approaching the patient.
* The Participant Information Sheet with info on the study shall be supplied to the patient by the research assistant and an opportunity shall be offered for any questions from the patient and their family/carers if appropriate, with the patients consent. Informed consent shall then be taken by a University of Strathclyde research assistant only.
* Participants will be supported to access and use the rehabilitation technology, in addition to usual care, by NHS staff. This will involve the prescription of a rehabilitation technology programme by the ward NHS physiotherapists, occupational therapists and speech and language therapists, following usual care assessment. This is with an aim to increase rehabilitation activity within the participant's capacity, taking into account their level of impairment and fatigue. Therefore, time spent using the rehabilitation technology will be varied and tailored to meet the participant's needs. The dose and intensity of technology enriched rehabilitation will be measured and recorded, however will not be controlled for these reasons.
* The Principal Investigator (NHS occupational therapist) will hold weekly meetings with the ward therapy staff to discuss any concerns around the study or regarding participant programs and will liaise directly with the research assistant as appropriate.
* Data collection/outcome measures will be completed as follows; Measures of recruitment and adherence Levels of recruitment (percentage of eligible individual consenting to participate) and attrition (percentage of people dropping/opting out before discharge) will be monitored and collated by the research assistant.

Duration spent on activities within the 'technology enriched rehabilitation space' will be timed by the NHS staff supporting the participants within the room, and these will be collated by the research assistant.

Additional outcome measures In order to further inform future studies the research team will collate the scores of the standard care

* Any Serious Adverse Effects (SAE) should be reported immediately to the Principal Investigator and a report made
* Participants' involvement in the study will end upon discharge from the stroke unit, or if withdrawn from the study for medical reasons or by personal choice.

Sample size Sample size / detectable difference. For a between-group difference of 1.6 points on the 15-point Rivermead Mobility Index (SD 3.0) (GAPS Study, Glasgow Augmented Physiotherapy Study (GAPS) group, 2004) with α = 0.05 and 80% power, the study requires ≈56 participants per group. Allowing for 10% attrition, the recruitment target of 62 participants per group is considered sufficient. The previous feasibility study recruited 60 participants over 9 months, a similar target is therefore regarded as achievable. A larger sample size for the virtual group (matched on diagnosis, age and Heath Board area) is planned (n=150) to improve statistical power. This would give a total sample of 212.

Data Analysis Analysis will be completed by the research team at the University of Strathclyde.

This pilot efficacy study will test the superiority of technology enriched rehabilitation over usual care by comparing the primary outcome measure (mRMI).

Exploratory analysis of other outcome measures of balance, upper limb function and walking recorded from the sample at UHW will be used to understand change in the primary variable (mRMI).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of new stroke by NHS Lanarkshire physician
* More than 48 hours since stroke event
* Deemed medically fit for rehabilitation by medical staff
* Deemed to require rehabilitation
* Able to provide informed consent

Exclusion Criteria:

* Acutely medically unwell
* Active cardiac disease, such as unstable angina
* Active delirium/significant levels of confusion
* Seizure within past 7 days
* Individual currently being managed under the Adults with Incapacity Act, unless the responsible medic has noted within the document that the individual has capacity to consent to rehabilitation research
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Modified Rivermead Mobility Index (MRMI) | Baseline (between consent and start of intervention) and immediately before hospital discharge.
  The Modified Rivermead Mobility Index (MRMI) is a standardized 8-item assessment that evaluates mobility tasks including turning over, balance, transfers, walking, and stair climbing. Scores range from 0 to 40, with higher scores indicating greater mobility. The items include:
  Turning over Lying to sitting Sitting balance Sitting to standing Standing Transfers Walking indoors Stairs

SECONDARY OUTCOMES:
10-Metre Walk Test (10MWT) | Baseline (between consent and start of intervention) and immediately before hospital discharge.
  A standardized assessment of gait speed over a 10-metre distance. Faster times indicate better walking ability.
Five Times Sit-to-Stand Test (FTSTST) | Baseline (between consent and start of intervention) and immediately before hospital discharge.
  A functional lower-limb strength and mobility test measuring the time required to stand up from a seated position five times. Shorter times indicate better performance.
Berg Balance Scale (BBS) | Baseline (between consent and start of intervention) and immediately before hospital discharge.
  A 14-item scale assessing static and dynamic balance. Scores range from 0 to 56, with higher scores indicating better balance.
Action Research Arm Test (ARAT) | Baseline (between consent and start of intervention) and immediately before hospital discharge.
  A standardized 19-item measure of upper-limb function assessing grasp, grip, pinch, and gross arm movement. Scores range from 0 to 57; higher scores indicate better arm function.
Grip Strength | Baseline (between consent and start of intervention) and immediately before hospital discharge.
  Maximum isometric grip force measured using a dynamometer. Higher values indicate greater strength.
Therapy Outcome Measure (TOM) | Baseline (between consent and start of intervention) and immediately before hospital discharge.
  A multidimensional clinical scale capturing impairment, activity, participation, and well-being
Fatigue Assessment Scale (FAS) | Baseline (between consent and start of intervention) and immediately before hospital discharge.
  A 10-item questionnaire evaluating physical and mental fatigue. Scores range from 10 to 50, with higher scores indicating more severe fatigue.
Length of Initial Hospital Stay | Through completion of the initial hospital stay.
  Total number of days from hospital admission to discharge.
Hospital Readmissions | Through study completion and up to 12 months post hospital discharge.
  Number of unplanned readmissions to any hospital setting.
Stroke Recurrence | Through study completion and up to 12 months post hospital discharge.
  Number of clinically confirmed recurrent strokes.
Prescription Use | Through study completion and up to 12 months post hospital discharge.
  Number and type of prescribed medications captured from medical records.
Ongoing Rehabilitation Use | Through study completion and up to 12 months post hospital discharge.
  Use (number of sessions) of outpatient or community-based rehabilitation services following discharge.
GP Visits | Through study completion and up to 12 months post hospital discharge.
  Number of visits to primary care providers during the follow-up period.
Level of Paid Social Care | Through study completion and up to 12 months post hospital discharge
  Amount and type of paid social care support used by participants (e.g., home care hours).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kerr, Study Director — Strathclyde; Gillian Sweeney, PhD, Principal Investigator — NHS Lanarkshire

IPD SHARING:
Plan to Share IPD: Yes
Data will be posted on the University's Data Sharing repository (PURE)
Supporting Information: Study Protocol, CSR
Time Frame: July 2027 Until July 2032
Access Criteria: This will be publicly available
URL: https://www.strath.ac.uk/research/researchdatamanagementsharing/datadeposit/

REFERENCES:
- [Result] Kerr A, Keogh M, Slachetka M, Grealy M, Rowe P. An Intensive Exercise Program Using a Technology-Enriched Rehabilitation Gym for the Recovery of Function in People With Chronic Stroke: Usability Study. JMIR Rehabil Assist Technol. 2023 Jul 21;10:e46619. doi: 10.2196/46619. PMID 37477954
- [Result] Sweeney G, Boyd F, Keogh M, Lyczba P, Forrest E, Rowe P, Barber M, Kerr A. A technology-enriched approach to increasing rehabilitation dose after stroke: Clinical feasibility study. Clin Rehabil. 2025 Jun;39(6):740-749. doi: 10.1177/02692155251333542. Epub 2025 Apr 18. PMID 40247700
- [Result] Gittins M, Vail A, Bowen A, Lugo-Palacios D, Paley L, Bray B, Gannon B, Tyson S. Factors influencing the amount of therapy received during inpatient stroke care: an analysis of data from the UK Sentinel Stroke National Audit Programme. Clin Rehabil. 2020 Jul;34(7):981-991. doi: 10.1177/0269215520927454. Epub 2020 Jun 7. PMID 32508132